CLINICAL TRIAL: NCT01209312
Title: Timing of Pre-meal Insulin Versus Accurate Carbohydrate Counting in Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-0931
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- full bolus -20 (Experimental): Will administer full insulin bolus 20 minutes prior to meal
  Interventions: Other: Bolus timing and dosing
- Full bolus, T0 (Experimental): Will administer full meal bolus at the start of the meal
  Interventions: Other: Bolus timing and dosing
- 1/2 bolus, T-20 (Experimental): Will only give half the insulin dose 20 minutes before meal
  Interventions: Other: Bolus timing and dosing
- 1/2 bolus T0 (Experimental): Will give half the amount of insulin at the time of the meal
  Interventions: Other: Bolus timing and dosing

INTERVENTIONS:
Other: Bolus timing and dosing — We will be altering the timing and dosages of the prescribed meal bolus.

SUMMARY:
The investigators are hoping to figure out how youth with type 1 diabetes can best control their blood glucose levels after meals, by determining whether accurate carbohydrate dosing or the timing of the bolus is more important. There is evidence to suggest that each strategy is important for blood glucose control. Unfortunately, for some people, prebolusing is difficult, because they may not know how much they are going to eat. To give an exact dose of insulin 20 minutes before a meal can be difficult. In this study, the investigators would like to show that taking even just part of the insulin bolus 20 minutes before the meal is preferable to waiting until mealtime and taking the entire bolus. To do this, the investigators will have 24 patients in the study, who will each spend 4 mornings at The investigators clinic. The order of the visits will be selected randomly. The visits will include: taking full bolus at mealtime, taking full bolus 20 minute before mealtime, taking ½ bolus at mealtime, and taking ½ bolus 20 minutes before mealtime. At each visit, the person will eat the same meal, but the timing and amount of the bolus will be different. The investigators will measure the blood glucose levels with a blood glucose meter, and also with a laboratory test called YSI. The investigators will also be measuring the glucose levels under the person's skin with a continuous glucose monitor. The investigators will compare the area under the curve for the different visits, as well as the glucose levels at different points after the meal.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-21, inclusive
* Diagnosis of type 1 diabetes for >1 year
* Using carbohydrate counting to dose mealtime insulin
* Using an insulin pump and continuous glucose monitor to control diabetes
* HbA1c <10%

Exclusion Criteria:

* Celiac disease or other GI abnormality
* Severe hypoglycemia in the past 6 months
* Pregnancy
* Documented hypoglycemia unawareness

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose area under the curve | 4 hours post-meal

CONTACTS AND LOCATIONS:
Overall Officials: H Peter Chase, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States